CLINICAL TRIAL: NCT03886948
Title: A Safety, Tolerability, and Pharmacokinetic Study of Injections of LY3074828 Solution Using Investigational 1-mL Pre-filled Syringes and Investigational 1-mL Autoinjector in Healthy Subjects
Brief Title: A Study of Injections of LY3074828 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16780; I6T-MC-AMBE (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-03-21; First posted 2019-03-22 (Actual); Results first posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 125 mg LY3074828 Prefilled Syringe (PFS) (Experimental): Reference 1: Participants received 125 mg LY3074828 solution formulation subcutaneously (SC) via 1-mL pre-filled syringe (PFS) administered in the arm.
  Reference 2: Participants received 125 mg LY3074828 solution formulation SC via 1-mL PFS administered in the thigh.
  Reference 3: Participants received 125 mg LY3074828 solution formulation SC via 1-mL PFS administered in the abdomen.
  Interventions: Drug: LY3074828; Device: Pre-filled syringe (PFS)
- 125 mg LY3074828 Autoinjector (AI) (Experimental): Test 1: Participants received 125 mg LY3074828 solution formulation SC via 1-mL Autoinjector (AI) administered in the arm.
  Test 2: Participants received 125 mg LY3074828 solution formulation SC via 1-mL AI administered in the thigh.
  Test 3: Participants received 125 mg LY3074828 solution formulation SC via 1-mL AI administered in the abdomen.
  Interventions: Drug: LY3074828; Device: Autoinjector (AI)

INTERVENTIONS:
Drug: LY3074828 — Administered subcutaneously (SC)
Device: Pre-filled syringe (PFS) — PFS used to administer LY3074828
  Arms: 125 mg LY3074828 Prefilled Syringe (PFS)
Device: Autoinjector (AI) — AI used to administer LY3074828
  Arms: 125 mg LY3074828 Autoinjector (AI)

SUMMARY:
The purpose of this study is to learn about the effects of LY3074828 when given as an injection just under the skin by two different devices. The study will last about 12 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

- Must be healthy males or females

Exclusion Criteria:

* Must not have an average weekly alcohol intake that exceeds 21 units/week (males) and 14 units/week (females)
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 8 weeks of screening, or intend to during the study
* Must not have been treated with steroids within 1 month of screening, or intend to during the study
* Must not be immunocompromised
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to Day 1
* Must not have significant allergies to humanised monoclonal antibodies
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test 1: 125 mg LY3074828: Participants received 125 mg LY3074828 solution formulation subcutaneously (SC) via 1-mL Autoinjector (AI) administered in the arm.
- Test 2: 125 mg LY3074828: Participants received 125 mg LY3074828 solution formulation SC via 1-mL AI administered in the thigh.
- Test 3: 125 mg LY3074828: Participants received 125 mg LY3074828 solution formulation SC via 1-mL AI administered in the abdomen.
- Reference 1: 125 mg LY3074828: Participants received 125 mg LY3074828 solution formulation SC via 1-mL pre-filled syringe (PFS) administered in the arm.
- Reference 2: 125 mg LY3074828: Participants received 125 mg LY3074828 solution formulation SC via 1-mL PFS administered in the thigh.
- Reference 3: 125 mg LY3074828: Participants received 125 mg LY3074828 solution formulation SC via 1-mL PFS administered in the abdomen.
Period: Overall Study
Arm/Group | Test 1: 125 mg LY3074828 | Test 2: 125 mg LY3074828 | Test 3: 125 mg LY3074828 | Reference 1: 125 mg LY3074828 | Reference 2: 125 mg LY3074828 | Reference 3: 125 mg LY3074828
Started | 11 | 11 | 11 | 11 | 11 | 11
Received at Least One Dose of Study Drug | 11 | 11 | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Test 1: 125 mg LY3074828 | Test 2: 125 mg LY3074828 | Test 3: 125 mg LY3074828 | Reference 1: 125 mg LY3074828 | Reference 2: 125 mg LY3074828 | Reference 3: 125 mg LY3074828 | Total
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (12.9) | 35.8 (11.5) | 44.8 (11.7) | 37.3 (15.2) | 41.3 (11.8) | 43.5 (10.8) | 40.7 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 5 | 6 | 6 | 36
  Male | 4 | 5 | 5 | 6 | 5 | 5 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 5 | 4 | 3 | 3 | 21
  Not Hispanic or Latino | 9 | 7 | 6 | 7 | 8 | 8 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 2 | 1 | 2 | 2 | 3 | 14
  White | 6 | 9 | 10 | 7 | 8 | 8 | 48
  More than one race | 1 | 0 | 0 | 1 | 1 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 11 | 11 | 11 | 11 | 66

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3074828
Description: Pharmacokinetics (PK): Maximum Observed Drug Concentration (Cmax) of LY3074828
Time Frame: Day 1: 0, 2, 6 hours, Day 2: 24 hours, Day 4, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85
Population: All participants who received at least one dose of study drug and had evaluable PK data. Per protocol, PK analysis were performed to evaluate solution formulation using a 1-mL PFS and a 1-mL AI.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: microgram/milliliter (ug/mL)
Groups:
- 125 mg LY3074828 AI: Participants received 125 mg LY3074828 solution formulation SC via 1-mL AI administered in the arm, thigh or abdomen.
- 125 mg LY3074828 PFS: Participants received 125 mg LY3074828 solution formulation SC via 1-mL PFS administered in the arm, thigh or abdomen.
Arm/Group | 125 mg LY3074828 AI | 125 mg LY3074828 PFS
Number analyzed (Participants) | 33 | 33
microgram/milliliter (ug/mL) | 9.19 (44) | 8.19 (56)

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Time t (AUC(0-tlast) of LY3074828, Where t is the Last Sample With a Measurable Concentration
Description: PK: Area Under the Concentration Versus Time Curve from Time Zero to Time t (AUC(0-tlast) of LY3074828, where t is the Last Sample with a Measurable Concentration
Time Frame: Day 1: 0, 2, 6 hours, Day 2: 24 hours, Day 4, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: microgram*day/milliliter (ug*day/mL)
Arm/Group | 125 mg LY3074828 AI | 125 mg LY3074828 PFS
Number analyzed (Participants) | 33 | 33
microgram*day/milliliter (ug*day/mL) | 146 (39) | 130 (51)

3. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC[0-∞]) of LY3074828
Description: PK: Area Under the Concentration Versus Time Curve from Time Zero to Infinity (AUC[0-∞]) of LY3074828
Time Frame: Day 1: 0, 2, 6 hours, Day 2: 24 hours, Day 4, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85
Population: All participants who received at least one dose of study drug and had evaluable PK data. Per protocol, PK analysis were performed to evaluate formulation using a 1-mL PFS and a 1-mL AI.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: ug*day/mL
Arm/Group | 125 mg LY3074828 AI | 125 mg LY3074828 PFS
Number analyzed (Participants) | 33 | 33
ug*day/mL | 149 (38) | 133 (50)

4. Primary Outcome: Visual Analog Scale (VAS) Pain Score by Device
Description: The pain VAS is a participant-administered single-item scale designed to measure pain using a 0-100 millimeter (mm) horizontal VAS. Overall severity of participant's pain is indicated by placing a single mark on the horizontal 100 mm scale from 0 mm (no pain) to 100 mm (severe pain).
Time Frame: Day 1: 1, 5 (±1.5) and 15 (±2) minutes
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | 125 mg LY3074828 AI | 125 mg LY3074828 PFS
Number analyzed (Participants) | 33 | 33
millimeter (mm)
  1 Minute | 27.2 (25.0) | 22.9 (21.5)
  5 Minutes (±1.5) | 8.3 (14.3) | 10.9 (15.5)
  15 Minute (±2) | 2.3 (5.8) | 2.8 (6.3)

5. Primary Outcome: Visual Analog Scale (VAS) Pain Score by Device and Injection Site Location
Description: as for outcome 4
Time Frame: Day 1: 1, 5 (±1.5) and 15 (±2) minutes
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Test 1: 125 mg LY3074828 | Test 2: 125 mg LY3074828 | Test 3: 125 mg LY3074828 | Reference 1: 125 mg LY3074828 | Reference 2: 125 mg LY3074828 | Reference 3: 125 mg LY3074828
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11
millimeter (mm)
  1 Minute | 30.1 (24.9) | 27.4 (30.5) | 24.1 (20.9) | 26.7 (23.5) | 22.5 (25.6) | 19.5 (15.5)
  5 Minutes (±1.5) | 6.5 (9.8) | 12.2 (22.0) | 6.4 (7.1) | 11.8 (20.1) | 8.9 (13.7) | 11.9 (13.2)
  15 Minutes (±2) | 1.8 (2.9) | 3.8 (9.5) | 1.4 (2.5) | 3.6 (10.1) | 1.7 (2.0) | 3.1 (4.4)

ADVERSE EVENTS:
Time Frame: Up To 85 Days
Description: All participants who received at least one dose of study drug.
Arm/Group | Test 1: 125 mg LY3074828 | Test 2: 125 mg LY3074828 | Test 3: 125 mg LY3074828 | Reference 1: 125 mg LY3074828 | Reference 2: 125 mg LY3074828 | Reference 3: 125 mg LY3074828
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 3/11 | 2/11 | 2/11 | 1/11 | 2/11 | 7/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1: 125 mg LY3074828 (N=11) | Test 2: 125 mg LY3074828 (N=11) | Test 3: 125 mg LY3074828 (N=11) | Reference 1: 125 mg LY3074828 (N=11) | Reference 2: 125 mg LY3074828 (N=11) | Reference 3: 125 mg LY3074828 (N=11)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-17): https://cdn.clinicaltrials.gov/large-docs/48/NCT03886948/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-04): https://cdn.clinicaltrials.gov/large-docs/48/NCT03886948/SAP_001.pdf